CLINICAL TRIAL: NCT02719041
Title: Predictive Biomarkers for IGF1R Targeted Therapy in Ovarian Cancer: a Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-19-16
Record Dates: First submitted 2016-03-13; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Tissue samples: Tissue samples taken from women treated for ovarian cancer will be stained.
  Interventions: Other: Immunohistochemistry staining method

INTERVENTIONS:
Other: Immunohistochemistry staining method

SUMMARY:
The main goal of this study is to employ a novel proteomic approach to identify predictive tumor biomarkers that will increase the efficacy of insulin-like growth factor (IGF1R) targeted therapy in epithelial ovarian cancer. It is expected that these predictive biomarkers will be applied to increase the response rate in selected groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* women who underwent surgery for ovarian cancer

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The tissue and medical history of forty women who underwent surgery for ovarian cancer, at the Hillel Yaffe Medical Center
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Responsive to IGF1R therapy | One year
  Mean tumor volume will be calculated and growth inhibition will be reported as the percentage decrease of tumor volume compared with the control.

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Bruchim, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No